CLINICAL TRIAL: NCT07382323
Title: Transdiagnostic Metacognitive Therapy Compared to Disorder-specific Cognitive-behavioral Therapy for Anxiety Disorders: a Qualitative Study
Brief Title: Metacognitive Therapy Compared to Cognitive-behavioral Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KI-2025-07875-02
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder; Social Anxiety Disorder; Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdiagnostic metacognitive therapy (Experimental): Metacognitive therapy in a transdiagnostic format; a single treatment protocol is used for all three anxiety disorders
  Interventions: Behavioral: Transdiagnostic metacognitive therapy
- Disorder-specific cognitive-behavioral therapy (Active Comparator): Cognitive-behavioral therapy in a disorder-specific format; each of the three anxiety disorders is treated using a separate treatment protocol
  Interventions: Behavioral: Disorder-specific cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Transdiagnostic metacognitive therapy — Metacognitive therapy focuses on metacognitions.
  Arms: Transdiagnostic metacognitive therapy
Behavioral: Disorder-specific cognitive-behavioral therapy — Cognitive-behavioral therapy focuses on cognitions and/or behaviors.
  Arms: Disorder-specific cognitive-behavioral therapy

SUMMARY:
This is a qualitative study of participants who have taken part in a randomized controlled trial comparing transdiagnostic metacognitive therapy and disorder-specific cognitive-behavioral therapy for anxiety disorders. The purpose of the study is to explore participant perceptions of the respective treatment models to facilitate implementation and dissemination of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* A principal diagnosis of generalized anxiety disorder, social anxiety disorder, or posttraumatic stress disorder,
* No change in dose during the last six weeks if on pharmacological treatment, and
* Ability to read and speak Swedish.

Exclusion Criteria:

* A current diagnosis of psychotic disorder, bipolar disorder, neurocognitive disorder, or moderate to severe substance use disorder,
* Acute suicide risk, or
* Concurrent psychological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative interview data | Up to 13 weeks
  Participant responses based on questions posed in an interview

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
The datasets analyzed in this study are not publicly available due to legal and ethical restrictions under Swedish data protection regulations. Requests for access may be directed to the Data Protection Officer at Stockholm Health Care Services, and are subject to approval by the relevant data governance authorities. Requests to access the datasets should be directed to gdpr.slso@regionstockholm.se.